CLINICAL TRIAL: NCT06302751
Title: An Electronic Remote Application to Improve the Postoperative Outcomes in Colorectal Cancer Patients: Single-center, Interventional Study
Brief Title: A Mobile Application to Improve Postoperative Outcomes in Colorectal Cancer
Acronym: RAISe-Care
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3647
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Colorectal Cancer; Surgery
Keywords: Colorectal cancer; Surgery; Mobile app; Unplanned readmissions
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, interventional case-series study with a historical cohort of comparison
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Care 4 Today ® (Johnson and Johnson) mobile app (Experimental): Patients will undergo standard perioperative management. Additionally, patients will use the Care 4 Today ® (Johnson and Johnson) mobile app for remote monitoring from the preoperative assessment day to 30 days after surgery. The Care 4 Today Care ® (Johnson and Johnson) mobile app will include daily reminds for preoperative recommendations adherence (water intake, medications adherence, mobilization, smoking quit...) and postoperative monitoring of symptoms (fever, pain, and mood deflections).
  Interventions: Device: Care 4 Today ® (Johnson and Johnson) mobile app
- Standard perioperative management (No Intervention): The historic cohort include patients who underwent standard perioperative management from March 2020 to April 2023.

INTERVENTIONS:
Device: Care 4 Today ® (Johnson and Johnson) mobile app — Care 4 Today ® (Johnson and Johnson) mobile app will cover the perioperative period spanning through the preoperative assessment day (approximately -seven to -one from surgery) to 30 days after surgery and will monitor the adherence to preoperative and postoperative recommendations.
  Arms: Care 4 Today ® (Johnson and Johnson) mobile app

SUMMARY:
The unplanned readmission rate after colorectal cancer surgery is still high, despite the implementation of enhanced recovery programs. The use of a mobile-based application for perioperative remote monitoring may improve the postoperative outcomes and reduce the unplanned postoperative readmissions.

DETAILED DESCRIPTION:
Despite the implementation of enhanced recovery programs, the rate of unplanned readmissions remains high after colorectal cancer surgery. These readmissions are often preventable with a better postoperative management. Increasing studies have demonstrated the feasibility and efficacy of perioperative remote monitoring mobile applications in improving the postoperative outcomes but are often limited to one restricted outcome. This project aims to evaluate the effect of the Care 4 Today® (Johnson & Johnson) perioperative mobile app on the postoperative outcomes of colorectal cancer patients, with a focus on unplanned readmissions.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years old.
* Patients scheduled for elective curative colorectal resection, including right (or extended) colectomy, left colectomy, rectal resection (with or without ileostomy), total colectomy, recanalization, or multiple colon resection.
* Patients willing to comply with the study procedures.
* Proficient understanding of the Italian language

Exclusion Criteria:

* Any condition that, in the opinion of the investigator, may interfere with the study procedures.
* Patients scheduled for palliative surgery.
* Patients with a planned elective intervention requiring urgent or emergent surgery will be withdrawn from the study.
* Pregnant or breastfeeding women.
* Inability to comply with the study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Unplanned hospital readmissions | 30 days after surgery
  Rate difference of unplanned hospital readmissions between the experimental group and historical cohort of comparison.

SECONDARY OUTCOMES:
Severity of postoperative complications | 30 days after surgery
  Compare the severity of postoperative complications- classified according to the Clavien-Dindo scale (ranging from 0 [no postoperative complications] to 5 [postoperative complications leading to death]- between the experimental group and historical cohort of comparison.
Length of hospital stay | From the day of surgery to the day of discharge
  Compare the median length of hospital stay (calculated in days from the day of surgery to the day of discharge) between the experimental group and the historical cohort of comparison.
Time from symptoms onset to diagnosis | 30 days after surgery
  Compare the time (in hours) from symptoms onset to diagnosis of postoperative complications occurring in the experimental group and historical cohort of comparison.
Healthcare costs | 30 days after surgery
  Compare the healthcare resources utilization between the experimental group and the historical cohort of comparison.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Foppa, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan; Spinelli Antonino, MD, PhD, Principal Investigator — Humanitas Research Hospital IRCCS, Rozzano-Milan
Locations (1):
- IRCCS Humanitas Research Hospital, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No